CLINICAL TRIAL: NCT06864273
Title: Increasing Access to Hearing Healthcare: An Assessment of Pharmacy Technician Educational Training for the Provision of Over-the-Counter Hearing Aids in Rural Alabama and Mississippi Pharmacies
Brief Title: Assessing Pharmacy Technician Educational Training for the Provision of Over-the-Counter Hearing Aids in Rural Alabama and Mississippi Pharmacies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pittsburgh (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A24-0556; R21DC022070 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Bilateral Hearing Loss; Health Services Research
Keywords: pharmacy education; rural health; Aids, Hearing
MeSH Terms: conditions — Hearing Loss, Bilateral; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The educational pharmacy technician training includes four sequential stages. Each technician will receive stepped interventions of "No Training", followed by "Online Modules," then "Online Discussions and Assigned Readings," and finish with "Practicum." The practicum experience will involve providing over-the-counter hearing aids to adults with bilateral mild-to-moderate hearing loss. Once completed, pharmacy technicians will have experienced a multimodal form of educational training that is considered best practices by the American Society of Health System Pharmacists and the Accreditation Council for Pharmacy Education for training pharmacy technicians, which must include didactic, simulated and experiential training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alabama and Mississippi Pharmacy Technicians (Experimental): Pharmacy technicians from Alabama and Mississippi will progress through four different steps of educational training for the purpose of assisting with the provision of over-the-counter hearing aids in rural Alabama and Mississippi counties. The types of training include four weeks of no training (control condition), four weeks of viewing online modules, four weeks of participating in online discussions, and four weeks of practical experiences. The practicum will include using hearing screening equipment to help assess hearing loss in adults, and setting over-the-counter hearing aid controls for adults with mild-to-moderate hearing bilateral hearing loss.
  Interventions: Behavioral: Pharmacy Technician Educational Training

INTERVENTIONS:
Behavioral: Pharmacy Technician Educational Training — Pharmacy Technicians will participate in a stepped-wedge educational training program. The first step will be a control condition where they will receive no training, the second step will include viewing online modules, the third step will include online discussions, and the fourth step will include practical experiences with adults with bilateral hearing loss. Pre-training quizzes and surveys will be completed before and after each step.

SUMMARY:
Hearing loss is a major public health concern due to its negative association with emotional well-being, cognition, and physical ailments, such as diabetes. Access to audiologists and otolaryngologists in many regions across the US is poor or extremely limited. Rural populations are older, less educated, and have lower household incomes compared to populations in metropolitan areas. Also, with increasing age adults experience greater rates of hearing loss. Fortunately, the 2022 FDA Final Rule for Over-the-Counter Hearing Aids (OTC HAs) could revolutionize assess to hearing aids and hearing healthcare by allowing adults with perceived mild-to-moderate hearing loss to purchase these devices over the counter, without medical clearance or care from an audiologist. Pharmacies located in rural areas now have the option to provide OTC HAs, something previously not possible. Currently, however, there are no established guidelines for effective provision of these devices in pharmacies located in rural communities. Educating pharmacy technicians to provide basic hearing healthcare related to OTC HAs use could address a critical need and create a new care delivery model to ensure sustainable, long-term access to hearing healthcare. The long-term goal of this study is to create a sustainable interprofessional collaborative between audiologists and pharmacists for the development of a hearing healthcare model that improves access and affordability of care in rural regions across the country. The specific aims are to 1) Determine an effective approach for educating pharmacy technicians for the provision of OTC HAs in rural community pharmacies, and 2) Identify satisfaction of care provided by pharmacy technicians and initial performance with OTC HAs in adults with hearing loss living in rural communities. A stepped wedged clinical trial design will be used to study the effectiveness of a comprehensive educational training program for pharmacy technicians. Technicians from rural Alabama and Mississippi, placed within four different clusters, will participate in a multimodal training program for the purpose of developing basic clinical skills to assist adults with perceived mild-to-moderate hearing loss. Additionally, adults with hearing loss who receive clinical services from trained pharmacy technicians will be asked to report on the care they received and benefit from their OTC HAs. The central hypotheses are a) that pharmacy technician training will result in greater understanding of hearing healthcare concepts compared to no training, and b) the training will lead to successful provision of basic hearing healthcare to adults with hearing loss in rural communities. The expected outcome of this project will be the establishment of a multimodal education program, leveraging the increased access of OTC HAs, to support those with hearing loss in rural pharmacies across the county. The ability of pharmacy technicians to provide this support will dramatically increase the availability of hearing services in rural communities, which will positively impact the quality of life for those with hearing loss.

DETAILED DESCRIPTION:
Many adults with hearing loss have no access to hearing healthcare due to a variety of factors1. One primary factor is that approximately 56% of counties across the US have no available audiological services. These counties are characterized by lower household incomes and older populations. Within some of these rural communities in Alabama, Hay-McCutcheon and colleagues found that adults with hearing loss did not know where to obtain services, travel distance to an audiologist was excessive, finances or insurance was lacking, some denied having hearing loss, and many did not know how to begin to address a hearing loss. Not addressing a hearing loss has significant implications for emotional well-being and mental health. Studies have found that hearing loss is associated with increased social isolation and loneliness. These conditions, in turn, can lead to cognitive decline. In addition to mental health, hearing loss has been associated with diabetes, affecting physical well-being. Considering the impact that hearing loss can have on general well-being, it is imperative that new models of care are developed to address this public health concern, especially for those living in rural and underserved communities, where access to hearing healthcare is limited. Addressing access to hearing healthcare for rural and underserved communities is a primary goal outlined in the 2016 National Academies of Sciences, Engineering, and Medicine document, Hearing Health Care for Adults: Priorities for Improving Access and Affordability10 and within the Notice of Special Interest for this application, Hearing Healthcare for Adults: Improving Access and Affordability (NOT-DC-21-001).

In an attempt to address the lack of hearing healthcare for adults, the FDA issued a Final Rule for OTC HAs in 2022. This rule allows adults who are 18 years of age or older with perceived mild-to-moderate hearing loss to purchase OTC aids without a medical exam, from an unlicensed seller, and without a prescription or fitting from an audiologist. Consequently, many adults without access to hearing healthcare now have the option to address their own hearing loss. Currently, these hearing aids can be purchased from retail stores, pharmacies, or online, and can range from approximately $200 per pair to up to $3000 per pair. However, for those who do not have geographical access to retail outlets, the internet, or who are not technologically astute, these potential solutions to hearing loss will remain elusive. Large retail chains are not easily accessible in rural communities, nor is access to the internet. To mitigate this problem, new care delivery models are needed to assist those with hearing loss across racial, educational, and economic lines. The study outlined in this proposal, where pharmacy technicians will be trained to assist rural populations with the provision of OTC HAs, is significant because it will be the first step for the development of a new care delivery model to increase access of hearing healthcare. Within the audiology field, it is not uncommon for support staff to be trained to assist with hearing assessments, such as newborn hearing screenings, elder care in hospitals, and hearing screenings for elementary school children. Educating technicians to assist pharmacists with the provision of OTC HAs, therefore, is a logical step to address hearing healthcare.

In rural communities, the pharmacy provides support to residents in a variety of ways. Pharmacists are trusted professionals who are trained to care for their patients and their medication-related needs. Community pharmacies have been referred to as untapped resources for public health. The pharmacy profession supports expanding roles for pharmacy technicians. Literature has suggested that their roles should be expanded to provide more point-of-care treatment, such as cholesterol and blood glucose screening, increasing duties associated with the technical aspects of pharmacy operations, and pharmacy administration duties. The development of a new care delivery model where the professions of audiology and pharmacy can work together to increase access to hearing healthcare in rural communities is highly significant.

Results from rigorous clinical trials conducted by Humes and colleagues in a largely white, highly educated, metropolitan college community demonstrated that adults with hearing loss can effectively set consumer driven (CD), or OTC, hearing aids independently. But data from these studies also suggested that adults were more satisfied with the hearing aids if they were given help setting the device. Over the past two years we have been conducting a clinical trial with OTC HAs (ID: NCT04671381) in West Central and South Alabama and unpublished preliminary data from 29 participants on a measure of hearing handicap found a large Cohen's d effect size of 0.91 when comparing adults who received no guidance setting their OTC HAs to those who received guidance after four weeks of OTC HA use. These data further stress the importance of developing care delivery models for rural communities to assist with the provision of OTC HAs.

Information from this study will provide the basis for interprofessional collaboration among audiologists, pharmacists, and pharmacy technicians for the provision of basic hearing healthcare in rural communities with older and poor populations. Also, the study will identify best practices for educating pharmacy technicians in the provision of OTC HAs in rural and communities. Importantly, these contributions will address an area of need outlined in the Hearing Healthcare for Adults: Improving Access and Affordability (NOT-DC-21-001), which is to increase access to hearing healthcare in diverse populations using innovative care delivery models.

ELIGIBILITY:
Inclusion Criteria:

1. Pharmacy technicians licensed to practice in the state of Alabama or Mississippi.
2. Pharmacy technicians who practice in rural communities of Alabama and Mississippi.
3. Adults 18 years of age with mild to moderate hearing loss and who live in rural communities of Alabama or Mississippi.

Exclusion Criteria:

1. Pharmacy technicians with hearing loss who could have prior understanding of care for those with hearing loss will not be included in the study.
2. Adults 18 years of age or older with typical hearing will not be included in the study.
3. Adults with hearing loss who live in urban areas of Alabama and Mississippi will not be included in the study.
4. Participants will be excluded if they have any medical condition resulting in cognitive impairment that results in an inability to complete the study tasks (e.g., mental health condition, stroke, head injury, dementia, or Alzheimer's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pre- and Post-training Quiz | From enrollment to the end of the educational training at 16 weeks.
  This quiz will assess knowledge and skills that are provided in during the 16-weeks of educational training that pharmacy technicians will receive. It will be administered before and after each training step.
Pre- and Post-training Confidence in Skills | From enrollment to the end of the educational training at 16 weeks.
  The questions in this survey will assess confidence levels of pharmacy technicians in assisting adults with hearing loss who receive over-the-counter hearing aids in their community pharmacy. It will be administered before and after each training step.

SECONDARY OUTCOMES:
Training Satisfaction Survey | From enrollment to the end of the educational training at 16 weeks.
  This survey will be completed by pharmacy technicians. Questions will assess how satisfied these participants are with the educational training they receive. It will be completed before and after each of the four training steps.
Satisfaction of Care Survey | This survey will be completed by adults with hearing loss at the end of the 4 weeks of the pharmacy technician practicum.
  This survey will assess how satisfied adults with hearing loss are with the care provided to them by a pharmacy technician.
Use and Care for Hearing Aids Survey | This survey will be completed by adults with hearing loss at the end of the 4 weeks of pharmacy technician practicum.
  This survey will be completed by adults with hearing loss who receive over-the-counter hearing aids from pharmacy technicians. It will assess how frequently they use their hearing aids and how they care for them.
Revised Hearing Handicap Inventory (RHHI) | This survey will be completed by adults with hearing loss at enrollment and at the end of the 4 weeks of hearing aid use.
  This 18-question survey measures emotional and social/situational consequences of hearing loss. It will be completed by adults before they receive over-the-counter hearing aids from pharmacy technicians. It will be repeated at the end of 4-weeks of hearing aid use.
International Outcome Inventory for Hearing Aids (IOI-HA) | This survey will be completed by adults with hearing loss prior to receiving hearingthe end of the 4 weeks of hearing aid use.
  The IOI-HA computes hearing aid benefit by calculating the difference between aided and unaided conditions. This survey will be completed by adults with hearing loss before they receive their over-the-counter hearing aids from the pharmacy technician. It will also be completed after 4-weeks of hearing aid use.
Abbreviated Profile of Hearing Aid Benefit (APHAB) | This survey will be completed by adults with hearing loss prior to receiving hearing aids and at the end of 4 weeks of hearing aid use.
  With this established survey, adults will report the benefit they receive from their over-the-counter hearing aids. It will compute hearing aid benefit by calculating the difference between aided and unaided conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia J Hay-McCutcheon, PhD, Principal Investigator — The University of Alabama; Lucas Berenbrok, PharmD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - The Department of Communicative Disorders, Box 870242, Tuscaloosa, Alabama
  - The Department of Communicative Disorders, Tuscaloosa, Alabama

IPD SHARING:
Plan to Share IPD: Yes
All raw data generated from surveys, including demographic data, and other scientific data, will be preserved and shared. Participant identifiers will not be shared.
Supporting Information: ICF, CSR
Time Frame: Release of a complete data set will to the Inter-university Consortium for Political and Social Research (ICPSR) occur within 12 months of the end of project data collection. Data used for the generation of manuscripts will be shared prior to publication. Data stored with the Data Sharing for Demographic Research (DSDR) repository through ICPSR will be available to the research community in perpetuity.
Access Criteria: For Public Use Data, all deidentified data that is not designated as restricted use data will be made publicly available via DSDR. To use these data, researchers must register with ICPSR and agree to the terms of use, which are designed to protect study participants. The sharing or redistribution of data downloads is not allowed. Datasets in DSDR are identified using a study digital object identifier (DOI), created by ICPSR. The DOI will allow researchers to find and identify data.
URL: https://www.openicpsr.org/openicpsr/project/221462/version/V1/view

REFERENCES:
- [Background] Brothers EB, Hay-McCutcheon MJ, Hughes PJ, Friend ML. Audiology, Medicine, and Pharmacy Interprofessional Preliminary Interviews and Discussions: Improving Hearing Health Care in Rural Alabama. Am J Audiol. 2022 Sep;31(3):656-668. doi: 10.1044/2022_AJA-21-00272. Epub 2022 Jun 23. PMID 35737896
- Available data/document: Informed Consent Form — https://www.openicpsr.org/openicpsr/ — Informed consent document can also be directly requested from the Principal Investigator, Marcia Hay-McCutcheon at mhaymccu@ua.edu